Relationship Between Acute Phase Markers and Post-operative Pain in Open Tension-free Inguinal Hernia Repair: An Observational Study

May 3, 2023

**Background**: Many patients undergoing Open Tension-free Inguinal Hernia Repair are prone to developing acute and chronic post-operative pain.

The aim of the study is to show a possible correlation between pain and acute phase proteins in order to:

- predict the severity of pain;
- select most suitable pain relief therapy for the patient.

**Materials and methods**: The day after surgery, some serum markers are determined by a blood sample. The markers analyzed are:

- Leukocytes;
- C-reactive protein (CRP);
- D-dimer;
- Fibrinogen;
- Neutrophil-to-Lymphocyte Ratio (NLR).

Pain level is assessed using the NRS scale at different times:

- 1st post-operative day;
- 7th post-operative day;
- One month after surgery;
- Three months after surgery;
- Six months after surgery.

Other data collected for the study are: gender, age and BMI.

**SAP**: Statistical Analysis Plan was expressed as percentages, median, and range of values. Differences between continuous variables were analyzed with the Mann-Whitney U test, whereas differences between categorical variables were evaluated with the chisquare or the Fisher's exact test, when appropriate. Variables achieving statistical significance (P<0.05) at univariate analysis were entered in a backward multivariate logistic regression model, removing the variable if P more than 0.10. P less than 0.05 was considered statistically significant. Statistical analysis was carried out with the SPSS software packaging (SPSS Inc., Chicago, IL), version 13.

## References

- 1. Hill AD, Banwell PE, Darzi A, Menzies-Gow N, Monson JR, Guillou PJ. Inflammatory markers following laparoscopic and open hernia repair. Surg Endosc. 1995 Jun;9(6):695-8. doi: 10.1007/BF00187942. PMID: 7482166.
- 2. Kokotovic D, Burcharth J, Helgstrand F, Gögenur I. Systemic inflammatory response after hernia repair: a systematic review. Langenbecks Arch Surg. 2017 Nov;402(7):1023-1037. doi: 10.1007/s00423-017-1618-1. Epub 2017 Aug 22. PMID: 28831565.
- 3. Vats M, Pandey D, Saha S, Talwar N, Saurabh G, Andley M, Kumar A. Assessment of systemic inflammatory response after total extraperitoneal repair and Lichtenstein repair for inguinal hernia. Hernia. 2017 Feb;21(1):65-71. doi: 10.1007/s10029-016-1543-1. Epub 2016 Nov 12. PMID: 27838831.
- 4. Choi HR, Song IA, Oh TK, Jeon YT. Perioperative C-reactive protein is associated with pain outcomes after major laparoscopic abdominal surgery: a retrospective analysis. J Pain Res. 2019 Mar 27;12:1041-1051. doi: 10.2147/JPR.S187249. PMID: 31114292; PMCID: PMC6497830.
- 5. Tarasov DA, Lychagin AV, Yavorovkiy AG, Lipina MM, Tarasova IA. C-reactive protein as marker of post-operative analgesic quality after primary total knee

- arthroplasty. Int Orthop. 2020 Sep;44(9):1727-1735. doi: 10.1007/s00264-020-04551-8. Epub 2020 Apr 16. PMID: 32300831.
- 6. Esme H, Kesli R, Apiliogullari B, Duran FM, Yoldas B. Effects of flurbiprofen on CRP, TNF-α, IL-6, and postoperative pain of thoracotomy. Int J Med Sci. 2011 Mar 10;8(3):216-21. doi: 10.7150/ijms.8.216. PMID: 21448308; PMCID: PMC3065790.
- 7. Rathee A, Chaurasia MK, Singh MK, Singh V, Kaushal D. Relationship Between Pre- and Post-Operative C-Reactive Protein (CRP), Neutrophil-to-Lymphocyte Ratio (NLR), and Platelet-to-Lymphocyte Ratio (PLR) With Post-Operative Pain After Total Hip and Knee Arthroplasty: An Observational Study. Cureus. 2023 Aug 20;15(8):e43782. doi: 10.7759/cureus.43782. eCollection 2023 Aug. PubMed ID: 37731439
- 8. Shu B, Xu F, Zheng X, Zhang Y, Liu Q, Li S, Chen J, Chen Y, Huang H, Duan G. Change in perioperative neutrophil-lymphocyte ratio as a potential predictive biomarker for chronic postsurgical pain and quality of life: an ambispective observational cohort study. Front Immunol. 2023 Apr 12;14:1177285. doi: 10.3389/fimmu.2023.1177285. eCollection 2023. PubMed ID: 37122722
- 9. Gonzalez-Callejas C, Aparicio VA, De Teresa C, Nestares T. Association of Body Mass Index and Serum Markers of Tissue Damage with Postoperative Pain. The Role of Lactate Dehydrogenase for Postoperative Pain Prediction. Pain Med. 2020 Aug 1;21(8):1636-1643. doi: 10.1093/pm/pnz325. PubMed ID: 31845982